CLINICAL TRIAL: NCT07133386
Title: TRUST Trial Protocol
Brief Title: TRicuspid Uk STudy
Acronym: TRUST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 338776
Record Dates: First submitted 2025-08-19; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Multicentre, blinded, placebo-controlled randomised clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-TEER arm (Experimental): Interventional device delivered via the transferral venous route to improve computation of the tricuspid valve leaflets with the aim of reducing tricuspid regurgitation.
  Interventions: Device: transcatheter edge to edge repair
- Placebo (Placebo Comparator): no therapeutic intervention undertaken. Patient will have all the same steps as the TriClip arm without actually having the TriClip device or delivery system inserted into the body.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: transcatheter edge to edge repair — Implantation of a tricuspid transcatheter edge to edge device
  Arms: T-TEER arm
Device: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a multicentre, randomised, placebo-controlled trial conducted at St Bartholomew's Hospital, John Radcliff Hospital, Royal Brompton Hospital, and Kings College London Hospital. The aim is to evaluate the benefits in health status from transcatheter edge to edge repair with the TriClip device in patients with severe or more symptomatic tricuspid regurgitation. A total of 150 patients will be recruited in a 1:1 ratio for TriClip or placebo. The primary endpoint of this study (change in Kansas City Cardiomyopathy Questionnaire between the treatment and placebo arm) will be analysed using a linear mixed model and compared between patients who receive the TriClip versus those who have a placebo procedure.

Study duration: 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years at recruitment
* Severe or more symptomatic TR determined by transthoracic echocardiography
* Optimized medical and/or device therapy for a minimum of 30 days
* Medications, including diuretics should be stable over the past 30 days
* Baseline KCCQ 75 or less on minimum 2 assessments at least 2 weeks apart
* New York Heart Association (NYHA) Functional Class II or ambulatory class IV
* Morphology of tricuspid valve suitable for TEER with expectation of a reduction of severity of TR to moderate or less
* Willing to provide written informed consent

Exclusion Criteria:

* Presence of anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results or result in an expected life expectancy of less than 12 months
* Active malignancy associated with a prognosis of <1 year
* Left ventricular ejection fraction (LVEF)<20%
* Tricuspid valve leaflet anatomy which may preclude TriClip implantation, proper clip positioning on the leaflets or sufficient reduction in TR. This may include:

  * Evidence of calcification in the grasping area
  * Presence of a severe coaptation defect (>10mm) of the tricuspid leaflets. - Severe leaflet defect(s) preventing proper device placement
  * Ebstein Anomaly - Identified by having a normal annulus position while the valve leaflets are attached to the walls and septum of the right ventricle.
* Tricuspid valve anatomy not evaluable by transthoracic (TTE) or transoesophageal echo (TOE)
* Rheumatic heart disease affecting the tricuspid valve
* Indication for left-sided (e.g. severe aortic stenosis, severe mitral regurgitation) or pulmonary valve correction. Note: Patients with concomitant mitral and tricuspid valve disease will have the option of having any significant mitral regurgitation managed, then waiting 60 days prior to being reassessed for the current trial.
* Pacemaker or implantable cardioverter-defibrillator (ICD) leads that would prevent appropriate placement of the TriClip.
* Tricuspid valve stenosis - Defined as a tricuspid valve orifice of ≤ 3.0 cm2 and/or mean gradient ≥3 mmHg as measured by the transthoracic echocardiography
* Pregnant
* Unable to comply with study protocol
* Uncontrolled systemic hypertension with a systolic blood pressure >180mmHg or diastolic blood pressure >110mmHg
* Severe pulmonary hypertension (sPAP>70mmHg) or fixed pre-capillary pulmonary hypertension assessed by cardiac catheterization
* Stroke within prior 90 days
* Chronic dialysis
* Bleeding disorders or hypercoagulable state
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Ongoing infection requiring current antibiotic therapy (if temporary illness, patients may enrol 30 days after discontinuation of antibiotics with no active infection).
* Known allergy or hypersensitivity to device materials
* Evidence of intracardiac, inferior vena cava (IVC), or femoral venous mass, thrombus or vegetation.
* Enrolment in another clinical trial that involves treatment of tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | every 2 weeks twice before the intervention and for 3 months post-intervention
  health status questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided